CLINICAL TRIAL: NCT04080089
Title: Establishment of a Diagnosis and Treatment System for Information Processing Damage in Children With Obstructive Sleep Apnea Hypopnea Syndrome
Brief Title: Establishment of a Diagnosis and Treatment System for Information Processing Damage in Children With OSAHS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2018-06-220
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Surgical Procedures, Operative; Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Children over the age of 6 who came to the outpatient clinic of our hospital received the informed consent of the parents, and then included in the case group, conducted a self-made sleep questionnaire, established a file, and monitored the sleep on the Mofeh Time Sleep Apnea Monitor. The results were uploaded to the cloud system for analysis. 50 children with OSAHS were screened. Voluntary participation in the study; ability to complete all tests as well as magnetic resonance studies. Exclusion criteria: 1 mental retardation, generalized developmental disorders, severe physical and endocrine diseases, neurological diseases and other mental disorders; 2 visual and auditory diseases affecting the processing of cognitive information. 3 Psychiatric drugs were used in January.
  Interventions: Combination Product: Surgical treatment, drug therapy, remote cognitive training
- Control group: Children in the same age group of children with health checkups were screened for sleep and questionnaires without sleep. After receiving parental informed consent, 30 children were included in the control group. Exclusion criteria: 1 mental retardation, generalized developmental disorder, learning disabilities, conduct Disorders, severe physical and endocrine diseases, neurological diseases and other mental illnesses. 2 There are visual and auditory diseases that affect the processing of cognitive information.

INTERVENTIONS:
Combination Product: Surgical treatment, drug therapy, remote cognitive training — Surgical treatment：Children with OSAHS who had surgical indications and informed consent from the parents underwent tonsillectomy and adenoidectomy.
  drug therapy：For children whose parents only agree to receive medical treatment, montelukast sodium tablets are given for 6 months to reduce the inflammatory response of adenoids, tonsils, etc.
  remote cognitive training:For children whose parents did not agree to undergo surgery or medication, the cognitive function was evaluated at the time of enrollment, and cognitive training was performed. Individualized training programs were developed according to the cognitive assessment system, and cognitive function was evaluated again after one course of treatment.
  Groups: Case group

SUMMARY:
Obstructive sleep apnea hypopnea syndrome (OSAHS) is a common childhood sleep disorder with an incidence of 3% . Studies have confirmed that OSAHS can cause multiple systemic dysfunction in children, especially affecting cognitive function . Cognitive function is an important part of human advanced neurological activities, including neurobehavioral functions such as orientation, attention, concentration, alertness, behavior, execution, etc., as well as intelligence and verbal functions such as memory, learning, calculation, language, understanding, judgment, and logic. Reasoning and many other aspects. Impaired cognitive function often means poor academic performance, which is the most concern of parents. However, due to the limitations of cognitive assessment tools, most studies only conduct qualitative research on children's cognition, lack of quantitative research. . The underlying reason is that these studies lack the guidance of systematic intellectual theory and the support of cognitive quantitative assessment tools. At present, no one at home and abroad has systematically and comprehensively studied the cognitive impairment caused by OSAHS based on the most advanced cognitive theory.

Modern cognitive science believes that cognition, including human memory, decision, reasoning, classification, and planning, is an ability that can be added to "the treatment may change." Some skill and intelligence of human beings at a certain level of cognitive activity can be trained in the execution of certain practices and in the completion of a plan. Scenes, situational features, and tasks, whether material or symbolic, play an important role in human training techniques.

Therefore, evaluable and scientific cognitive function training for individuals is beneficial to the development of cognitive function, especially for the treatment training of patients with cognitive dysfunction. At present, the treatment of OSAHS is mainly for the treatment of primary disease such as oropharyngeal surgery, CPAP, etc. These treatments

DETAILED DESCRIPTION:
There are many differences between children's OSAHS and adult OSAHS. Children's OSAHS mainly causes cognitive and neuropsychological disorders, hyperactivity disorder, attention deficit hyperactivity disorder, aggressive behavior, learning decline and nocturnal enuresis. At present, there are many studies on cognitive impairment in children with OSAHS at home and abroad. Cognitive impairment mainly affects attention, memory, especially executive function, such as problem solving, planning, goal-oriented behavior and so on. Lau EY et al assessed cognitive function by Wechner intelligence scale, children's auditory task, digital vigilance test and so on. It was found that compared with the normal group, the language working memory of OSAHS children was significantly impaired . Peng Wanda et al used routine craniocerebral MRI sequence and fluid attenuated inversion recovery (FIAIR) sequence perpendicular to bilateral hippocampus for imaging. According to Scheltens standard and Fukudas method, the severity of (PVH), which was associated with hippocampal volume atrophy and white matter lesion, was evaluated. The changes of cognitive function were evaluated by Montreal Cognitive Assessment scale (MoCA) and Mini Mental State scale (MMSE). The results showed that hippocampal volume atrophy and white matter lesions were closely related to cognitive impairment in patients with OSAHS. Craniocerebral MRI technique can provide objective imaging basis for the diagnosis of cognitive impairment in patients with OSAHS . However, these studies also have shortcomings. first of all, most studies do not study the cognitive process of OSAHS children as a complete system, but only study the correlation between one side (subsystem) or some aspects of children's cognition. Such as memory, executive function and so on. Modern cognitive neuroscience holds that cognitive process is the process of receiving, coding, storing, extracting and using information in the brain, that is, the process of information processing. Whether OSAHS children have defects in the process of information processing has not been reported at home and abroad. Secondly, due to the limitations of cognitive assessment tools, there is a lack of quantitative research. Adenoidectomy (adenotonsillectomy,AT) is recognized as the most commonly used treatment for OSAHS . AT treatment can effectively relieve respiratory tract obstruction caused by the proliferation of lymphoid tissue in the upper airway during sleep. In recent years, it has been found that the inflammatory response mediated by 1eukotriene (LTS) plays an important role in the pathogenesis and progress of OSAHS. It has also been found that long-term continuous positive airway pressure ventilation (Continuous Positive Airway Pressure,CPAP) can reduce serum inflammation and improve cognitive impairment in children with OSAHS . These treatments relieve obstruction of the upper airway in children with OSAHS, relieve nocturnal hypoxia exposure, and help improve damaged cognitive function, but fully restore advanced brain function. That is, in the process of understanding objective things, the acquisition, coding, operation, extraction and use of sensory input information need to improve their cognitive function and cognitive skills through cognitive training.

However, DN-CAS is a system established by English background. If the system is introduced directly, it may not adapt to the Chinese background. For example, Chinese phonetic training, Chinese character dyslexia training, planning process training based on Chinese cultural background and so on may not be applicable, so it is necessary to improve and introduce Chinese background based on PASS theory.

The existing cognitive training systems at home and abroad can not form an electronic prescription system which can cooperate with the diagnostic results. The prescription form is presented in the traditional paper form and lacks good confidentiality, ease of use and storage management. The training system also lacks flexible support for personalized training of patients. Patients are under the guidance of the doctor on the spot, in the hospital venue to complete the training, the training process needs the doctor to carry on the artificial treatment and guidance. It is difficult for doctors to easily customize different training prescriptions for different patients, and it is also difficult to carry out the electronic management of patient training data. The existing cognitive training systems are stand-alone systems, and there is no integrated system of screening, diagnosis and training. The scope and effect of application are greatly limited, far from being able to meet the growing needs of patients. The training plan based on PASS theory should be a personalized scheme based on common principles to adapt to individuals with different cognitive function levels. Therefore, the system generates personalized electronic prescriptions according to the training knowledge base, in which different training levels, contents and processes are customized according to the level and characteristics of individual cognitive function. The electronic prescription is provided to the patient in an encrypted storage medium, and the patient uses it to carry out training at the telemedicine terminal. During the training, the electronic prescription can automatically guide the patients to carry out the training steps without artificial treatment and show the personalized training scene for the patients. The training process and results are automatically monitored and recorded to the training centre server for evaluation and analysis by doctors.

The computer cloud system to be developed in this project is mainly composed of electronic scale evaluation system and brain cognitive function monitoring system. The electronic scale evaluation system is a semi-quantitative computer cloud system for self-evaluation of clinical symptoms and physician-assisted clinical syndrome evaluation. Its working principle is that the computer takes the place of doctors to conduct directional consultation with patients. The results of consultation were transformed into semi-quantitative data and compared with the established mathematical models to provide doctors with semi-quantitative decision-making data. The advantage of the system is that because the computer performs semi-quantitative consultation instead of the doctor, the patient's current history, past history, general situation and symptoms can be collected in detail and semi-quantitatively. At the same time, the working time of the doctor is saved and the intensity of the doctor's work is reduced at the same time, to the greatest extent, the omission of consultation in the consultation of the doctor is avoided, and the working time of the doctor is saved at the same time. (2) because the semi-quantitative results are compared with the previous data models, doctors can find diseases in more case models and help doctors find quantitative evidence for qualitative diagnosis. (3) due to the detailed consultation of the computer, sense of security, which brings high quality services to patients and detailed medical services, has increased the compliance of diagnosis and treatment. The brain cognitive function detection system is a computer cloud system laboratory, which is composed of several brain cognitive function detection subsystems, which reflects the function of brain information and function. The system presents the target task composed of the simplest visual basic geometry through the display screen, enables the detection object to complete the target task by operating the computer, and records the accuracy and time of completion. By comparing the results with the established mathematical models, we can measure the information plus function in 16 aspects of the human brain. Due to the introduction of time and space as the evaluation index of brain cognitive function, the detection of brain cognitive function gets rid of the traditional scale evaluation and enters the level of objective evaluation of physics.

In summary, based on the international advanced cognitive science PASS theory, this project intends to establish a digital remote DN:CAS cognitive evaluation and training (DN:CAS) computer remote system under the Chinese background. The information processing process of OSAHS children was quantitatively evaluated, on the basis of which the classification of defects in children's OSAHS information processing process was further discussed, and a cognitive prescription and remote training system with independent intellectual property rights was constructed. Finally, a complete screening-diagnosis-training-reevaluation process based on cloud computing is formed, in order to provide a basis for personalized clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

Case group - Children over 6 years old who have snoring in our outpatient clinic Control group - Children in the same age group of children with health checkups, screened by sleep questionnaire and sleep monitoring without OSAHS

Exclusion Criteria:

Case group - 1 mental retardation, extensive developmental disorders, severe physical and endocrine diseases, neurological diseases and other mental disorders; 2 there are visual and auditory diseases affecting the processing of cognitive information. 3 Psychiatric drugs have been used in the past 1 month.

Control group -1 mental retardation, generalized developmental disorders, learning disabilities, conduct disorders, severe physical and endocrine diseases, neurological diseases and other mental illnesses. 2 There are visual and auditory diseases that affect the processing of cognitive information.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Case group: Children（>6years old）who have snoring will be included in the case group after receiving informed consent from the parents. A sleep questionnaire will be conducted. The results were uploaded for analysis and 50 children with OSAHS were screened. Voluntary participation in the study; ability to complete all tests as well as magnetic resonance studies. Exclusion criteria: 1 mental retardation, generalized developmental disorders, severe physical and endocrine diseases, neurological diseases and other mental disorders; 2 visual and auditory diseases affecting the processing of cognitive information. 3 used psychiatric drugs in the past 1 month Control group: 30 Healthy children in the same age group, without OSAHS, received parental informed consent.Exclusion criteria: Same
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluating information processing | 6 months
  Different treatments were chosen to treat patients with OSAHS. After treatment, the digital remote DNCAS cognitive evaluation system was used to evaluate the information processing process of the child. Compare with pre-treatment and explore whether there is a difference in the treatment effect of each treatment method on children with different subtypes of information processing.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Cai, M.D., Study Chair — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- SAHWenzhouMU, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided